CLINICAL TRIAL: NCT05782582
Title: Chronic Coronary Syndrome in Swedish Primary Care
Acronym: COSPRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Staffan Nilsson, General practitioner, associate professor, principal investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-04416-01; RÖ-961940 (Other Grant/Funding Number: ALF Grants Region, Östergötland)
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Primary Health Care; Diagnostic Imaging; Myocardial Perfusion Imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial. All of 47 primary health care centres in Region Östergötland are invited to take part. After acceptance the actual number of primary health care centres will be randomly allocated to to either package or standard investigation group. The aim is to include about 20 primary health care centers in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Package investigation (Experimental): 1. Resting ECG,
  2. Evaluation of risk according to PTP-table.
  3. Echocardiography,
  4. Exercise stress bicycle test (secondarily drug provocation) with injection of isotope for myocardial scintigraphy,
  5. Scanning for myocardial perfusion
  6. CAC-scoring with CT
  Interventions: Diagnostic Test: Package investigation; Device: Sound registration with Cadscore® and added risk calculation
- Standard investigation (Active Comparator): 1. Resting ECG
  2. Evaluation of risk according to PTP-table.
  3. Echocardiography.
  4. Exercise stress bicycle test.
  If judged to be needed according to clinical indication sequentially completed by:
  Echocardiography, Exercise stress bicycle test (secondarily drug provocation) with injection of isotope for myocardial scintigraphy and/or Coronary CTA. In addition, cardiac examinations done with other modalities chosen on clinical grounds will be examined in the study.
  ,
  Interventions: Diagnostic Test: Standard investigation

INTERVENTIONS:
Diagnostic Test: Package investigation — Investigations performed on a single visit, according to arm description
  Arms: Package investigation
Device: Sound registration with Cadscore® and added risk calculation — Recording of cardiac diastolic sounds enabling the calculation of a risk score.
  Arms: Package investigation
Diagnostic Test: Standard investigation — Sequential investigations according to arm description
  Arms: Standard investigation

SUMMARY:
The goal of this clinical trial is to learn about a new procedure for investigation of possible coronary heart disease and to see if it is faster, cheaper or more expensive, promotes healthier behavior, mental well-being, adherence to drugs for heart protection and the risk for cardiac events like acute myocardial infarction over years to come. The novelty in the procedure is that a myocardial perfusion scan to assess blood flow to areas of the heart muscle, echocardiography i.e., heart ultrasound and heart CT scan comes as a "package investigation" performed on the same day. According to existing routines, "standard investigation" an exercise stress bicycle test is done, as well as an echocardiography and if needed the work up is completed by a myocardial perfusion scan. The main questions the trial aims to answer are:

* are the results from the procedure given to the patient faster with package investigation as compared to standard investigation?
* does the cost differ between the package and standard investigation group?
* does self-reported physical activity, physical fitness, dietary habits and mental well-being differ between the package and standard investigation group at start and after one, three and five years?
* does prescription of drugs taken for heart protection and adherence to the prescribed drugs differ between the package and standard investigation group after two and five years?
* does the risk for heart events like acute heart infarction differ between package and standard investigation after two and five years?

Primary health care centers in Region Östergötland are randomly assigned to use either the new or existing procedure for investigation of possible coronary heart disease a so called cluster randomization. Patients who consult a physician at any of these primary health care centers are potential participants in the trial and are informed about the trial by written information, as they get their appointment for the medical investigation at either of two hospitals in the Region Östergötland. When the patient comes to the hospital for the investigations, he or she is asked to give written consent to the research i.e., to answer questionnaires now after one, three and five years, to let the researchers take part of the medical records, investigational results and data from medical registries over time.

DETAILED DESCRIPTION:
In primary health care patients with chest symptoms are common. In many cases the cause is benign but chronic coronary artery disease (CAD) must often be considered. In the clinical work, evaluation of symptoms and risk factors are fundamental for a plausible working diagnosis and to judge if any further investigation is needed. The probability of CAD for a person of a certain age, sex and character of chest symptoms, scored from 0-3, i.e. pretest probability (PTP) for CAD, is substantially lower now than it was a decade ago in western countries. Consequently, recent European guidelines recommend that further investigation to rule out CAD may be omitted if the risk for CAD is judged to be low (PTP<15 %) and there are no further cardiovascular risk factors. If further investigation is needed in the low-risk group, computed tomography angiography (CTA) is preferable. When the risk for CAD is judged to be intermediate (PTP> 15 %) an imaging investigation is advocated instead of the well-established exercise stress bicycle test. A much-used imaging test is myocardial perfusion scan in which an exercise stress bicycle test is performed, with the addition of an intravenous injection of a small amount of radioactive tracer, whereafter the myocardial blood flow is demonstrated by imaging. Sensitivity for myocardial perfusion scan to detect significant CAD is 87 % (95 % CI 83-90) in comparison with exercise stress bicycle test where it is only 58 % (95 % CI 46-69). Specificity is 70 % (95 % CI 63-76) and 62 (95 % CI 54-69) respectively. However, the exercise stress bicycle test reveals indirect signs of myocardial ischemia and is reasonable in price, easy to perform and available in many clinics and hospitals. It is since long the first-line method for referral from the primary care setting. If the result from the exercise stress bicycle test is inconclusive, the work-up should be continued, e.g. with myocardial perfusion scan. An echocardiogram is often performed as well to evaluate the condition of the myocardium, heart valves and left ventricular ejection fraction. This stepwise or sequential clinical work-up strategy is well known and reasonable in general practice where patients in general have a low prevalence of serious diseases compared to organ specialist clinics. Since June 2021 in Region Östergötland (471 912 inhabitants 2022) CTA is recommended if further investigation is deemed necessary in patients with a low risk of CAD (PTP< 15 %) in primary care. For patients with intermediate risk of CAD (PTP> 15 %) exercise stress bicycle test is still the first-line choice.

There may be advantages if myocardial perfusion scan and echocardiogram is performed on a single visit. In addition, a CT scan of the heart to determine coronary artery calcification (CAC) score is easy to perform on the same visit, gives only a small amount of radiation and adds useful information. The CAC-score has been shown to be an independent predictor of future cardiovascular events and is useful for reclassification of cardiovascular risk based on traditional risk factors like age, cholesterol levels and smoking habits. Furthermore, a clear and coherent answer on all three investigations, to the referring GP can provide a more secure basis for clinical decision making. For the individual patient it is probably an advantage to get a thorough investigation done at one single visit and possibly a faster and more valid statement from the investigations by the GP. On the other hand, if many advanced investigations are done unnecessarily, expenses and exposure to radiation will increase unjustifiably. Possibly there is also a risk of medicalization and to create worries for future cardiovascular events communicating the CAC-score to people that has not asked for the information.

In order to get a faster and more complete basis for the evaluation of CAD in primary care patients with an intermediate (PTP> 15 %) risk the investigators created a package investigation comprised of myocardial perfusion scan, echocardiogram and CT scan of the heart on a single visit. The results from myocardial perfusion scan will be written according to national guidelines and communicated to the referring GP together with results from echocardiogram and CAC-scoring as a coherent answer. Moreover, registration of heart sounds followed by risk calculation by a technical device Cadscore® will be performed but only for scientific analyzes and not be given as a clinical answer.

In this study the investigators aim to compare the standard routine sequential investigation for detecting CAD with a single-visit package investigation.

ELIGIBILITY:
Inclusion Criteria:

• People who seek primary care for symptoms judged to be compatible with a medium probability (PTP> 15) for symptomatic chronic coronary artery disease.

Exclusion Criteria:

* Suspicion of acute coronary syndrome when care is sought.
* Previously diagnosed acute myocardial infarction
* Revascularization with PCI/CABG
* Proven reversible ischemia according to myocardial scintigraphy.
* Left Bundle Branch Block (LBBB).
* Ventricular pacemaker
* People whose meaning due to illness, mental disorder, weakened state of health or any other similar condition cannot be obtained, to be included in a research project.
* Insufficient understanding of spoken and written Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of days till completed assessment of myocardial ischemia | From the day of inclusion up to one year
  waiting time (days) after the results of package investigation or exercise stress bicycle test (standard investigation) are available at the primary health care center till invasive coronary angiography is done or results from completed non-invasive myocardial ischemia investigation is communicated to the participant (patient).

SECONDARY OUTCOMES:
Swedish crowns or other currency | From the day of inclusion and one year thereafter
  Costs for medical investigations, consultations and costs generated by participants loss of production and travel costs. Data will be gathered by review of the participants computerized medical records one year after the day of inclusion. Medical investigations will be sought in local medical registries.The participant will be asked if being a professional worker or not on the day of inclusion.
Health related quality of life | Up to five years
  Health related quality of life will be measured by EQ-5D-5L Swedish version (Devlin NJ et al., 2017)
Radiation per patient | One year
  millisievert (mSv)
Physical activity | Up to five years
  Physical activity will be measured by two categorical questions asking for level of physical activity (Olsson SJ et al., 2016)
Dietary habits | Up to five years
  Dietary habits will be measured by five categorical questions about consumption of fruit, vegetables, snacks and soft drinks during the last week. (Henriksson H et al., 2020)
Health and life quality | Up to five years
  Health and life quality will be measured by the Swedish RAND-36 A 36-item scale. (Ohlsson-Nevo E et al., 2021)
Heart focused anxiety | Up to five years
  Heart focused anxiety will be measured by the Cardiac Anxiety Questionnaire - CAQ An 18-item scale (Eifert et al., 2000)
Generalized anxiety | Up to five years
  Generalized anxiety will be measured by the Brief Measure for Assessing Generalized Anxiety Disorder - GAD-7 A seven item scale. (Spitzer et al., 2006)
Depression symptoms | Up to five years
  Depression symptoms will be measured by the Patient Health Questionnaire - PHQ-9 Maximum score 27 (Hansson et al., 2009)
Sleep quality | Up to five years
  Sleep quality will be measured by The Pittsburgh Sleep Quality Index - PSQI A 19-item scale which assesses sleep quality and disturbances over a 1-month time interval. (Buysse et al., 1989)
Physical fitnes | Up to five years
  Physical fitness will be measured by The International Fitness Scale - IFIS A 5-item scale (Ortega FB et al., 2011)
MACE | Up to five years
  Major adverse cardiovascular event - MACE Data will be gathered from national Swedish registries i.e. SWEDEHEART, the National Patient Register and Dödsorsaksregistret (The Cause of Death Register)
Compliance to cardioprotective drugs | Two years before and up to five years after inclusion.
  Data on prescribed and purchased drugs will be gathered from the National Prescribed Drug Register .

OTHER OUTCOMES:
Presence of pathological q-waves | On the day of inclusion
  Resting ECG
Reversible ischemia | On the day of inclusion
  ST-depression provoked by exercise
Alcohol consumption | Up to five years
  Alcohol consumption will be measured by the Alcohol Use Disorders Identification Test - AUDIT. Score range: 0-40. (WHO-publications 2001)
Smoking | Up to five years
  Smoking will be measured by the question 'Do you smoke?' (No, I have never smoked/No, I have quitted/Yes, occasionally/Yes, daily) and quantified by the number of cigarettes per day.
Dental health | Up to five years
  Dental health will be explored by a 5-item questionnaire constructed for the study
Number of days on sick leave | Time frame: From the day of inclusion and one year thereafter
  Data will be gathered by review of the participants computerized medical records one year after the day of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Iredahl, MD, PhD, Principal Investigator — IMH/Community Medicine/Linkoping university
Locations (3):
- Sweden (3):
  - Department of Clinical Physiology, Linköping University Hospital, Linköping, Linköping
  - Hjärthälsan Linköping AB, Linköping
  - Department of Clinical Physiology, Vrinnevi Hospital, Norrköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Hoorweg BB, Willemsen RT, Cleef LE, Boogaerts T, Buntinx F, Glatz JF, Dinant GJ. Frequency of chest pain in primary care, diagnostic tests performed and final diagnoses. Heart. 2017 Nov;103(21):1727-1732. doi: 10.1136/heartjnl-2016-310905. Epub 2017 Jun 20. PMID 28634285
- [Background] Knuuti J, Ballo H, Juarez-Orozco LE, Saraste A, Kolh P, Rutjes AWS, Juni P, Windecker S, Bax JJ, Wijns W. The performance of non-invasive tests to rule-in and rule-out significant coronary artery stenosis in patients with stable angina: a meta-analysis focused on post-test disease probability. Eur Heart J. 2018 Sep 14;39(35):3322-3330. doi: 10.1093/eurheartj/ehy267. PMID 29850808
- [Background] Juarez-Orozco LE, Saraste A, Capodanno D, Prescott E, Ballo H, Bax JJ, Wijns W, Knuuti J. Impact of a decreasing pre-test probability on the performance of diagnostic tests for coronary artery disease. Eur Heart J Cardiovasc Imaging. 2019 Nov 1;20(11):1198-1207. doi: 10.1093/ehjci/jez054. PMID 30982851
- [Background] Winther S, Nissen L, Schmidt SE, Westra JS, Rasmussen LD, Knudsen LL, Madsen LH, Kirk Johansen J, Larsen BS, Struijk JJ, Frost L, Holm NR, Christiansen EH, Botker HE, Bottcher M. Diagnostic performance of an acoustic-based system for coronary artery disease risk stratification. Heart. 2018 Jun;104(11):928-935. doi: 10.1136/heartjnl-2017-311944. Epub 2017 Nov 9. PMID 29122932
- [Background] Budoff MJ, Young R, Burke G, Jeffrey Carr J, Detrano RC, Folsom AR, Kronmal R, Lima JAC, Liu KJ, McClelland RL, Michos E, Post WS, Shea S, Watson KE, Wong ND. Ten-year association of coronary artery calcium with atherosclerotic cardiovascular disease (ASCVD) events: the multi-ethnic study of atherosclerosis (MESA). Eur Heart J. 2018 Jul 1;39(25):2401-2408. doi: 10.1093/eurheartj/ehy217. PMID 29688297
- [Background] Mitchell JD, Fergestrom N, Gage BF, Paisley R, Moon P, Novak E, Cheezum M, Shaw LJ, Villines TC. Impact of Statins on Cardiovascular Outcomes Following Coronary Artery Calcium Scoring. J Am Coll Cardiol. 2018 Dec 25;72(25):3233-3242. doi: 10.1016/j.jacc.2018.09.051. PMID 30409567
- [Background] Devlin NJ, Brooks R. EQ-5D and the EuroQol Group: Past, Present and Future. Appl Health Econ Health Policy. 2017 Apr;15(2):127-137. doi: 10.1007/s40258-017-0310-5. PMID 28194657
- [Background] Olsson SJ, Ekblom O, Andersson E, Borjesson M, Kallings LV. Categorical answer modes provide superior validity to open answers when asking for level of physical activity: A cross-sectional study. Scand J Public Health. 2016 Feb;44(1):70-6. doi: 10.1177/1403494815602830. Epub 2015 Sep 21. PMID 26392418
- [Background] Henriksson H, Alexandrou C, Henriksson P, Henstrom M, Bendtsen M, Thomas K, Mussener U, Nilsen P, Lof M. MINISTOP 2.0: a smartphone app integrated in primary child health care to promote healthy diet and physical activity behaviours and prevent obesity in preschool-aged children: protocol for a hybrid design effectiveness-implementation study. BMC Public Health. 2020 Nov 23;20(1):1756. doi: 10.1186/s12889-020-09808-w. PMID 33228572
- [Background] Ohlsson-Nevo E, Hiyoshi A, Noren P, Moller M, Karlsson J. The Swedish RAND-36: psychometric characteristics and reference data from the Mid-Swed Health Survey. J Patient Rep Outcomes. 2021 Aug 4;5(1):66. doi: 10.1186/s41687-021-00331-z. PMID 34347192
- [Background] Eifert GH, Thompson RN, Zvolensky MJ, Edwards K, Frazer NL, Haddad JW, Davig J. The cardiac anxiety questionnaire: development and preliminary validity. Behav Res Ther. 2000 Oct;38(10):1039-53. doi: 10.1016/s0005-7967(99)00132-1. PMID 11004742
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Hansson M, Chotai J, Nordstom A, Bodlund O. Comparison of two self-rating scales to detect depression: HADS and PHQ-9. Br J Gen Pract. 2009 Sep;59(566):e283-8. doi: 10.3399/bjgp09X454070. PMID 19761655
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Ortega FB, Ruiz JR, Espana-Romero V, Vicente-Rodriguez G, Martinez-Gomez D, Manios Y, Beghin L, Molnar D, Widhalm K, Moreno LA, Sjostrom M, Castillo MJ; HELENA study group. The International Fitness Scale (IFIS): usefulness of self-reported fitness in youth. Int J Epidemiol. 2011 Jun;40(3):701-11. doi: 10.1093/ije/dyr039. Epub 2011 Mar 24. PMID 21441238
- [Derived] Nilsson S, Gabro F, Stertman E, Bernfort L, Fredrikson M, Henriksson P, Johansson P, Kastbom L, Karner Kohler A, Loof J, Mourad G, Olsson E, Valladares C, Ostgren CJ, Sederholm Lawesson S, Engvall J, Iredahl F. Chronic cOronary Syndrome in Swedish PRImary care (COSPRI)-a study protocol for a 5-year cluster randomized controlled trial on a novel package versus standard investigation in patients with suspected chronic coronary syndrome referred from primary health care. Trials. 2025 Jun 21;26(1):215. doi: 10.1186/s13063-025-08911-w. PMID 40544312
- See also: SWEDEHEART — https://www.ucr.uu.se/swedeheart/
- See also: The National Patient Register — https://www.socialstyrelsen.se/en/statistics-and-data/registers/national-patient-register/
- See also: Dödsorsaksregistret (The Cause of Death Register) — https://www.socialstyrelsen.se/statistik-och-data/register/dodsorsaksregistret/
- See also: The National Prescribed Drug Register — https://www.socialstyrelsen.se/en/statistics-and-data/registers/national-prescribed-drug-register/

DOCUMENTS (2):
  • Study Protocol: Study Protocol COSPRI_Issue1.2 (2026-01-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT05782582/Prot_003.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT05782582/SAP_001.pdf